CLINICAL TRIAL: NCT03614884
Title: Developing and Testing the Effectiveness of a Novel Online Integrated Treatment for Problem Gambling and Tobacco Smoking: A Randomized Controlled Trial
Brief Title: Effectiveness of an Online Integrated Treatment for Problem Gambling and Tobacco Smoking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2018:088 (HS22037)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Gambling Disorder
Keywords: gambling; smoking; online intervention; Cognitive Behavioural Therapy; Motivational Interviewing; Randomized Controlled Trial
MeSH Terms: conditions — Gambling; Smoking

STUDY DESIGN:
Intervention Model Description: A two-arm randomized controlled trial (RCT) will be conducted to evaluate the proposed online intervention. Eligible participants will be randomized to either the online integrated gambling and smoking treatment condition, or the gambling only (i.e., control) condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gambling and Smoking Treatment (Experimental): Participants in this arm will be given access to the online integrated treatment for gambling and smoking.
  Interventions: Behavioral: Gambling and Smoking Treatment
- Gambling Only Treatment (Active Comparator): Participants in this arm will be given access to the online gambling only treatment.
  Interventions: Behavioral: Gambling only treatment

INTERVENTIONS:
Behavioral: Gambling and Smoking Treatment — The treatment condition will have access to 7 treatment modules on content surrounding both gambling and smoking behaviours. Participants will have 8-weeks to complete them. The content of all modules is derived from Cognitive Behavioural Therapy and Motivational Interviewing. Through module engagement, participants will identify goals related to gambling and smoking behaviours, learn strategies to cope with cravings and triggers, and learn how to prevent relapse. Participants will have immediate access to all modules, and it will be recommended that they work through the modules sequentially. Participants in this condition will also be provided with nicotine replacement therapy (NRT) in the form of nicotine patches to use for the duration of the study.
  Other Names: Online CBT and MI
  Arms: Gambling and Smoking Treatment
Behavioral: Gambling only treatment — The control condition will have access to 7 treatment modules on content surrounding gambling only. Participants will have 8-weeks to complete them. The content of all modules is derived from Cognitive Behavioural Therapy and Motivational Interviewing. Through module engagement, participants will identify goals related to gambling behaviours, learn strategies to cope with cravings and triggers, and learn how to prevent relapse. Participants will have immediate access to all modules, and it will be recommended that they work through the modules sequentially.
  Other Names: Online CBT and MI
  Arms: Gambling Only Treatment

SUMMARY:
Research has shown that problem gambling and tobacco smoking are highly comorbid. Problem gamblers who smoke tend to: have more severe gambling problems, experience stronger gambling urges, have other mental disorders, bet larger sums of money, spend more time in gambling activities, and have greater financial problems. Accordingly, it might be helpful to reduce your smoking as well, while you are trying to get a grip on your gambling.

Previous studies have treated gambling on its own or tobacco smoking on its own. To date, there has not been a treatment that has targeted treating both at the same time. Considering how often these conditions occur together, it is important to see if combining their treatment results in beneficial outcomes. In the current research, the researchers aim to design and test an online, self-help intervention for co-occurring problem gambling and tobacco smoking. It will draw on strategies from Cognitive Behavioural Therapy (CBT) and Motivational Interviewing (MI) - both which have been shown to be successful in treating problem gambling and tobacco smoking. These outcomes will be compared to a group that receives treatment for problem gambling only. This research will provide insight into a potential new intervention for treating two highly co-occurring conditions.

DETAILED DESCRIPTION:
The researchers are hoping to recruit 300 participants for this study. Half (150) of these individuals will receive the integrated treatment, where both gambling and smoking behaviours will be addressed. Those in the integrated group will be encouraged to use nicotine replacement therapy (NRT) in the form of nicotine patches. These patches will be provided to participants at the beginning of the intervention and will be encouraged to use for the duration of the 8-weeks. The the other half of the participants (150) will receive the problem gambling treatment only.

Once participants provided informed consent and are registered on the treatment website, they will be asked to complete a baseline assessment in order to determine eligibility. Eligible participants will be those that: are aged 19 years old+, have at least moderate levels of gambling, report current daily smoking, are fluent in English, have weekly internet access, and report at least moderate motivation to change gambling and/or smoking behaviours.

Once the link is available, participants will complete the online, self-help 8-week treatment. At the end of the program, they will complete the same brief questionnaires. Six months following the completion of the online program, they will complete the same series of brief questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* ages 19+
* problem gambling status based on reporting a score of > 3 on the Problem Gambling Severity Index
* reporting current daily smoking
* fluency in English
* have weekly Internet access
* report at least moderate motivation to change gambling and/or smoking behaviours

Exclusion Criteria:

* Those that are identified as "Higher" risk on the suicide screener
* self-reported engagement in other psychosocial treatments for problem gambling and/or smoking
* past-90 day psychosis or mania
* presence of a severe substance use disorder (SUD) (For alcohol, individuals with a score of > 20 on the Alcohol Use Disorder Identification Test (AUDIT) will be excluded from the study. For substance use, individuals with a score of > 5 on the Drug Abuse Screening Test-10 (DAST-10) will be excluded).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of days gambled | Participants will be assessed using the TLFB at three time points: at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Timeline Follow-Back (TLFB; Sobell & Sobell, 1992) - designed to assess the number of days gambled during a 30-day period. The TLFB has been shown to provide reliable and valid estimates of gambling behaviour, and is widely used in basic and treatment studies.
Change in money spent gambling | Participants will be assessed using the TLFB at three time points: at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  TLFB designed to assess money (in dollars) spent gambling during a 30-day period.
Change in time spent gambling | Participants will be assessed using the TLFB at three time points: at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  TLFB designed to assess the time spent gambling (in minutes) during a 30-day period.

SECONDARY OUTCOMES:
Gambling symptom assessment | Change in score from beginning of program (baseline T0) at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Brief self-report questionnaire with questions about gambling symptoms
Problem gambling severity | Change in score from beginning of program (baseline T0) at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Brief self-report questionnaire with questions about gambling severity
Cigarette use | Participants will be assessed using the TLFB at three time points: at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  TLFB designed to assess the number of cigarettes smoked during a 30-day period.
Point Prevalence for Abstinence | Percentage of people at baseline (T0),immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Percentage of participants who remained abstinent from smoking in the 30-days prior to each assessment
Nicotine dependence symptoms | Change in score from beginning of program (baseline T0) at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Brief self-report questionnaire with questions about nicotine dependence

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Keough, PhD, Principal Investigator — University of Manitoba; Michael Schaub, PhD, Principal Investigator — University of Zurich; Sherry H Stewart, PhD, Study Chair — Dalhousie University; David Hodgins, PhD, Study Chair — University of Calgary; James Mackillop, PhD, Study Chair — McMaster University; R. Michael Bagby, PhD, Study Chair — University of Toronto
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilevicius E, Single A, Baumgartner C, Bui V, Kempe T, Schaub MP, Stewart SH, MacKillop J, Hodgins DC, Wardell JD, O'Connor R, Read J, Hadjistavropoulos H, Sundstrom C, Keough MT. Developing and testing the effectiveness of a novel online integrated treatment for problem gambling and tobacco smoking: a protocol for an open-label randomized controlled trial. Trials. 2020 Nov 19;21(1):937. doi: 10.1186/s13063-020-04867-1. PMID 33213506